CLINICAL TRIAL: NCT07320118
Title: Cell Therapy for Osteoarthritis
Brief Title: Does Surgical Treatment of Cartilage Defects Prevent Osteoarthritis in Later Life?
Acronym: REACT
Status: Recruiting | Type: Observational
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Collaborators: Keele University (Other)
Responsible Party: Sponsor
Other Study IDs: RL1 418
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis (OA)
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ACI patiients: Patient must have had ACI surgery at least 10 months prior
- Non ACI Patients: Control group of patients who did not have ACI

SUMMARY:
Observational study to assess the effectiveness of cell therapy for the treatment of osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* ACI patients or patients receiving an alternative treatment

Exclusion Criteria:

* Anyone who does not meet the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients based in the United Kingdom treated at RJAH orthopaedic hospital
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2010-04-13 (Actual); Primary Completion 2030-01-12 (Estimated); Study Completion 2030-01-12 (Estimated)

PRIMARY OUTCOMES:
Cell Therapy Questionnaire | At least fifteen months post operation
  Cell Therapy Questionnaire CTQ

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - The Robert Jones and Agnes Hunt Orthopaedic Hospital, Oswestry
  - Robert Jones and Agnes Hunt Orthopaedic hospital, Oswestry